CLINICAL TRIAL: NCT04414813
Title: Clinical Study of Stereotactic Transplantation of Human Amniotic Epithelial Stem Cells (hAESCs) in the Treatment of Parkinson's Disease (PD)
Brief Title: Stereotactic Transplantation of hAESCs for Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2019（CR）-001
Record Dates: First submitted 2019-05-21; First posted 2020-06-04 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; stereotactic transplantation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study plans to recruit 3 patients who meet the criteria. 50 millions HAESCs will be transplanted to participants with PD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAESCs treatment (Experimental): 50 millions hAESCs are transplanted to participants with PD.
  Interventions: Biological: Human Amniotic Epithelial Stem Cells

INTERVENTIONS:
Biological: Human Amniotic Epithelial Stem Cells — Stereotactic transplantation of hAESCs for participants with PD.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of stereotactic transplantation of hAESCs for Parkinson's disease.

DETAILED DESCRIPTION:
The study plans to recruit 3 participants with Parkinson's disease . Using stereotactic technology, hAESCs will be accurately transplanted into the lateral ventricle. Therapeutic effectiveness and safety of hAESCs on PD will be evaluated. hAESCs are derived from placental amnion donated after cesarean section in healthy women. hAESCs is developed from the epiblast as early as 8 days after fertilization, recent reports indicate that hAESCs have some characteristics of neural stem cell. These cells are able to differentiate into dopaminergic neurons and secrete dopamine and various neurotrophic factors. These HAESCs could be seen as one of the best potential stem cell source for treating Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. 30-70 years old, with primary Parkinson's disease more than 5 years, male or female;
2. The "off-stage"Hohen and Yahr grade of Parkinson's disease is from 2 to 4; and the"off-stage"UPDRS score is 38-70, difference between two scores before treatment is less than 10% ;
3. The dosage of medicine is stable for more than 3 months;
4. Levodopa treatment was effective ;
5. Stable condition, good control of complications, no general anesthesia contraindications, no contraindications to stereotactic surgery and other conditions that interfere with clinical evaluation;
6. No abnormalities affecting cell transplantation were found through head MRI;
7. Patients shall be properly cared during treatment, and caregivers can provide assistance to the researcher if necessary.

Exclusion Criteria:

1. Atypical Parkinson's disease, such as Parkinson's syndrome, secondary Parkinson's disease;
2. Only having tremor syndrome;
3. Serious movement disorders and cannot complete any routine exercise tasks;
4. Symptoms of severe neurological deficits caused by other diseases;
5. Severe mental symptoms or dementia;
6. Patients are unwilling to cooperate or incapable of completing self-evaluation, and cannot complete the evaluator with the help of a doctor;
7. History of striatum or extrapyramidal surgery, including deep brain stimulation (DBS);
8. Ongoing treatment of apomorphine injecting ;
9. Coagulation disorders or ongoing anticoagulation therapy;
10. Women of childbearing age who do not take effective contraception;
11. Pregnant or lactation;
12. Patients who have participated in other clinical studies of drugs or medical devices within 3 months;
13. Botox toxin, phenol, subarachnoid injection of baclofen or interventional therapy for the treatment of dystonia or spasticity within 6 months;
14. History of seizures or taking prophylactic anti-epileptic drugs;
15. General anesthesia or stereotactic surgery contraindications, such as sleep apnea, chronic obstructive pulmonary disease;
16. Other circumstances judged by the investigator that may cause negative effect to the subject;
17. Alcohol or drug abuse;
18. Used diazepam within 3 months;
19. Severe cognitive impairment, depression, or behavioral disorder, defined as the Mini-Mental State Assessment Scale (MMSE) of less than 26 points, and the Hamilton Depression Rating Scale (HAMD) of greater than 35 points;
20. Chest CT shows active disease or tumor;
21. Currently suffering from or ever had a tumor other than cutaneous basal cell tumor and cervical carcinoma in situ;
22. The detection of HIV, hepatitis B virus(HBV), hepatitis C virus (HCV), syphilis and other infection indicators before surgery can not exclude HIV and syphilis infection;
23. Abnormal liver and kidney normal function tests in the laboratory, liver and kidney function is defined as Alanine aminotransferase（ALT）, Aspartate aminotransferase（AST） is less than 2.5 times the upper limit of normal, blood urea nitrogen (BUN) and Creatinine（Cr） are less than the upper limit of normal.
24. Other situations not suitable for enrollment judged by investigator

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with adverse event and serious adverse event | 12 months
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment. A serious adverse event is defined as an adverse event that meets at least one of the following serious criteria: • fatal • life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • congenital anomaly/birth defect • other significant medical hazard. Whether an adverse event was treatment-related (TRAE) or not was determined by investigator.

SECONDARY OUTCOMES:
Changes in Unified Parkinson's Disease Rating Scale (UPDRS) in ON and OFF state | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  UPDRS is used for evaluating the impairment and disability associated with Parkinson's Disease (PD). It consists of four sections: (1) Mentation, behavior, and mood; (2) Activities of daily living (ADLs); (3) Motor; and (4) Complications.
  The UPDRS score ranges from 0 to 199, with higher score indicating greater disability.
Changes in the Hoehn and Yahr scale | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  Hoehn and Yahr scale is used to provide a general estimate of clinical function of PD patients, combining functional deficits (disability) and objective signs (impairment). The Hoehn and Yahr score ranges from 0 to 5, with higher score indicating higher dysfunction of PD patients.
Changes in Parkinson's Disease Questionnaire (PDQ-39) | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  PDQ-39 provides the evidence of the quality of life of a PD patient. The higher the score, the lower the quality of life of PD patients.
Changes in the Schwab and England score | day 0, 1 month, 2 month, 3 month, 6 month, 9 month and 12 month.
  The Schwab and England scale develop a scale that describes the capacity of daily living shown by a PD patient. It measures the following three areas: dependence, abilities, and awareness. The Schwab and England scores range from 0% to 100%, with higher scores indicating greater healthy status.
Levodopa equivalent daily dose | day 0, 1 month, 2 month, 3 month, 4 month, 5 month, 6 month, 9 month and 12 month.
  Differences in daily dosage of levodopamine
Cranial doparmin transporter measured by positron emission tomography(PET)-magnetic resonance Imaging(MRI) | 4 month, 6 month
  Changes of cranial expression of dopamine transporter investigated by PET-MR
Glucose metabolism measured by 18F-Fluoro-2-deoxy-glucose (FDG) PET scan | 4 month, 6 month
  Changes in cranial glucose metabolism investigated by PET-MR
Differences in biochemical indicators of cerebrospinal fluid | day 0, 1 month, 2 month, 3 month, 4 month,5 month,6 month, 9 month and 12 month.
  Cerebrospinal fluid indicator tests include biochemical indicators and the following parameters: Dopamine (DA), high vanillic acid (HVA), 5-hydroxytryptamine (5-HT), 5-hydroxyindoleacetic acid (5-HIAA), norepinephrine (MHPG), α synuclein (α-synuclein), amyloid deposition (Aβ42), Tau protein (Tau) Protein, Neurofilament light (NF-L), and yKL-40 (YKL-40).

CONTACTS AND LOCATIONS:
Overall Officials: WU Jingwen, Dr, Principal Investigator — Shanghai East Hospital, China
Locations (1):
- WU Jingwen, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No